CLINICAL TRIAL: NCT00241345
Title: Randomized Trial of Preemptive Treatment With Oral Valganciclovir Compared With IV Ganciclovir for Cytomegalovirus Infection After Bone Marrow or Peripheral Blood Stem Cell Transplant
Brief Title: Trial of Preemptive Treatment With Oral Valganciclovir Compared With Intravenous (IV) Ganciclovir for Cytomegalovirus Infection After Bone Marrow or Peripheral Blood Stem Cell Transplant
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to low accrual
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04-0274
Record Dates: First submitted 2005-10-17; First posted 2005-10-18 (Estimated); Last update posted 2013-07-23 (Estimated); Status verified 2013-07

CONDITIONS: Cytomegalovirus Infections
Keywords: post transplant; Any patient receiving an allogeneic bone marrow or peripheral blood stem cell transplant at Washington University Medical Center
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — Valganciclovir; Ganciclovir

ARMS (2):
- Group A (Experimental): IV ganciclovir (5mg/kg every 12 hours for 7 days followed by 5mg/kg every 24 hours for 7 days. If CMV viral load <5000 copies/ml after 14 days then 5mg/kg every 24 hours for a total of 21 total days of therapy. If CMV viral load >5000/ml but less than index viral load after 14 days then 5mg/kg every 24 hours for a total of 28 total days of therapy. If CMV viral load >= index viral load after 14 days then 5mg/kg every 12 hours for 7 days. If repeat CMV viral load is <= the previous CMV viral load then 5mg/kg every 12 hours for an additional 7 days.
  Interventions: Drug: Ganciclovir
- Group B (Experimental): PO valganciclovir (900 mg every 12 hours for 7 days followed by 900 mg every 24 hours for 7 days. If CMV viral load <5000 copies/ml after 14 days then 900 mg every day until 21 total days of therapy. If CMV viral load >5000 copies/ml after 14 days but less than the index viral load then 900 mg every day until 28 total days of therapy. If CMV viral load >= the index viral load 900 mg every 12 hours for 7 days, if CMV viral load <= to previous viral load then 900 mg every 12 hours for another 7 days.
  Interventions: Drug: Valganciclovir

INTERVENTIONS:
Drug: Valganciclovir
  Arms: Group B
Drug: Ganciclovir
  Arms: Group A

SUMMARY:
The purpose of this trial is to determine if preemptive therapy with oral valganciclovir is as effective as intravenous ganciclovir in clearing cytomegalovirus (CMV) viremia as determined by quantitative CMV polymerase chain reaction (PCR) assay in patients who have undergone bone marrow or peripheral blood stem cell transplant.

DETAILED DESCRIPTION:
* To study the effect of preemptive therapy with IV ganciclovir and PO valganciclovir as determined by quantitative CMV PCR.
* To determine the incidence of CMV disease and CMV related mortality following preemptive treatment with oral valganciclovir and IV ganciclovir.
* To compare the incidence of recurrent CMV viremia after treatment with PO valganciclovir to that seen after treatment with IV ganciclovir.
* To determine the toxicity profile of valganciclovir.
* To screen for mutations in the UL97 gene in patients who have increasing CMV viral loads after 14 days of treatment.
* To determine if patients treated with PO valganciclovir have ganciclovir drug levels which are equivalent to those seen in historical control subjects treated with PO valganciclovir.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving allogeneic peripheral blood stem cell transplant from either a related or unrelated donor at Washington University Medical Center.
* An initial episode of CMV viremia.
* At the time of randomization:

  * ANC greater than or equal to 1000
  * Age greater than or equal to 18
  * Adequate renal function with creatinine clearance greater than 10 ml/min
  * Total bilirubin less than or equal to 3.0

Exclusion Criteria:

* Current GI graft versus host disease grade III-IV
* Development of CMV disease prior to or at the time of the first detection of CMV viremia by PCR
* Uncontrolled emesis or diarrhea (greater than or equal to 4 episodes per day) for 2 consecutive days
* Pregnant or nursing female patient
* Known hypersensitivity to ganciclovir

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2004-06; Primary Completion 2007-11 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
If preemptive therapy with oral valganciclovir is as effective as intravenous ganciclovir in clearing CMV viremia as determined by quantitative CMV PCR assay in patients who have undergone allogeneic bone marrow or peripheral stem cell transplant. | 4 weeks from start of therapy
  Clearance of CMV viremia will be defined as CMV viral load less than 5,000 copies/ml of whole blood.

SECONDARY OUTCOMES:
Effect of preemptive therapy with IV ganciclovir and PO valganciclovir as determined by quantitative CMV PCR. | 6 months
Incidence of CMV disease and CMV related mortality following preemptive treatment with oral valganciclovir and IV ganciclovir. | 6 months
Compare the incidence of recurrent CMV viremia after treatment with PO valganciclovir to that seen after treatment with IV ganciclovir. | 6 months
Toxicity profile of valganciclovir | 6 months
Mutations in the UL97 gene in patients who have increasing CMV viral loads after 14 days of treatment | 14 days
Determine if patients treated with PO valganciclovir have ganciclovir drug levels which are equivalent to those seen in historical control subjects treated with PO valganciclovir. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Vij, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu